CLINICAL TRIAL: NCT00840905
Title: A Pilot Observational Study to Determine the Prevalence of HPV Serology in HIV Seropositive Women From Subsaharan Africa and Brasil
Brief Title: A Study to Examine the Human Papillomavirus Types Exposure in Women From Southern Africa and Brasil
Status: Completed | Type: Observational
Sponsor: Cynthia S Firnhaber (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Cynthia S Firnhaber, Associate Professor of Medicine, University of Witwatersrand, South Africa
Organization: University of Witwatersrand, South Africa (Other)
Other Study IDs: Merck P0806
Record Dates: First submitted 2009-02-10; First posted 2009-02-11 (Estimated); Last update posted 2012-11-07 (Estimated); Status verified 2012-11

CONDITIONS: HIV; HIV Infections
Keywords: HPV
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: None Retained — Blood /plasma specimen 10cc
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: HIV seropositive women from an HIV Antiretroviral therapy clinic in Johannesburg South Africa
- 2: A cohort of HIV seropositive women from Gabarone Botswana
- 3: A cohort of HIV seropositive women from Rio De Janeiro Brasil

SUMMARY:
This is a study to determine what Human Papillomavirus HIV seropositive women in Botswana, South Africa and Brasil have been exposed to during their life. The Human Papillomavirus causes cervical cancer. Different types are more likely to lead to cancer than other types. A vaccine has been made to fight infection against HPV 16 and 18 which has been shown to cause cervical cancer in America and Europe. What HPV type cause cancer in other countries is not as well studied.

Hypothesis HPV serology will demonstrate that exposure to each HPV type in Gardisil (6,11,16,18) will be <50% in HIV seropositive women in resource limited countries.

DETAILED DESCRIPTION:
Plasma from HIV seropositive women will be taken and sent to MERCK in the USA to evaluate what the antibody titers of HPV 6,11,16 and 18. .

ELIGIBILITY:
Inclusion Criteria:

* HIV seropositive women 18 years of age and older Consent signed per local IRB requirement

Exclusion Criteria:

* Can not give blood

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV seropositive women from South Africa, Botswana, and Brasil
Sampling Method: Non-Probability Sample
Enrollment: 487 (Actual)
Dates: Start 2009-02; Primary Completion 2010-03 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To determine the seroprevalence of HPV types 6,11,16,18 in HIV serOpositive women for Botswana, South Africa and Brazil | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia S Firnhaber, MD, Principal Investigator — Clinical HIV Research Unit University of Witwatersrand
Locations (3):
- Shahin Lockman, Habarone, Botswana
- Fundacao Oswaldo Cruz, Rio de Janeiro, Brazil
- University of Witwatersrand/Helen Joseph Hospital, Johannesburg, South Africa